CLINICAL TRIAL: NCT07188194
Title: Prospective Value of Clinical , CSF and MRI Findings in Pediatric Acute Disseminated Encephalomyelitis
Brief Title: ADAM'S Prognostic Markers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa AboAlkasem Mohamed, Resident, Assiut University
Other Study IDs: ADAM'S prognostic markers
Record Dates: First submitted 2025-09-03; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Disseminated Encephalomyelitis
MeSH Terms: conditions — Encephalomyelitis, Acute Disseminated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children

SUMMARY:
Acute Disseminated Encephalomyelitis (ADEM) is an immune-mediated demyelinating disorder of the central nervous system that predominantly affects children. It typically presents with an acute onset of multifocal neurological symptoms, often preceded by a viral infection or, less commonly, vaccination. ADEM is characterized radiologically by widespread, bilateral, asymmetric lesions in the brain and spinal cord, and is often monophasic in nature.

Despite generally favorable outcomes, a subset of patients may experience significant neurological sequelae, prolonged recovery, or even conversion to chronic demyelinating disorders such as multiple sclerosis (MS) or multiphasic ADEM. The early identification of patients at risk for poor outcomes remains a clinical challenge, as the course of the disease is highly variable.

Cerebrospinal fluid (CSF) analysis and magnetic resonance imaging (MRI) are essential components in the diagnostic workup of ADEM. Certain CSF features-such as pleocytosis, elevated protein levels, or the presence of oligoclonal bands-may reflect the underlying immunological activity and CNS inflammation. Similarly, specific MRI characteristics-such as lesion distribution, size, contrast enhancement, or involvement of deep gray matter-may correlate with disease severity and long-term prognosis.

The clinical presentation of ADEM is heterogeneous. Common features include encephalopathy (ranging from irritability to coma), seizures, motor deficits, ataxia, visual disturbances, and brainstem symptoms. The severity and combination of these manifestations can vary widely between patients. Several studies suggest that certain clinical features may correlate with poorer prognosis, such as prolonged or deep coma, recurrent seizures, early need for intensive care, and delayed initiation of immunotherapy.

DETAILED DESCRIPTION:
* To evaluate the prognostic value of cerebrospinal fluid (CSF) and magnetic resonanceimaging (MRI) findings at initial presentation in predicting six months neurological outcomes in pediatric patients diagnosed with ADEM.
* Secondary aim : correlation between clinical presentation and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. - First episode of acute disseminated encephalomyelitis( ADEM).
2. - MRI and cerebrospinal fluid (CSF) performed within 7 days of symptom onset.
3. - Age from 6 months up to 18 years

Exclusion Criteria:

1. - History of prior demyelinating events
2. - Alternative diagnoses (e.g., CNS infections, metabolic disorders).

Ages: 6 Minutes to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 6 months -1 Year diagnosed with ADEM
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Neurological status assessed by the National Institutes of Health Stroke Scale (NIHSS) | At 3 months, and 6 months
  The NIHSS quantifies neurological impairment. Scores range from 0 (no deficit) to 42 (severe stroke). Higher scores indicate worse neurological status.

SECONDARY OUTCOMES:
Functional outcome assessed by the Modified Rankin Scale (mRS) | At 3 months and 6 months
  The mRS measures the degree of disability or dependence in daily activities. Scores range from 0 (no symptoms) to 6 (death). Higher scores indicate worse functional outcomes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anlar B, Basaran C, Kose G, Guven A, Haspolat S, Yakut A, Serdaroglu A, Senbil N, Tan H, Karaagaoglu E, Karli Oguz K. Acute disseminated encephalomyelitis in children: outcome and prognosis. Neuropediatrics. 2003 Aug;34(4):194-9. doi: 10.1055/s-2003-42208. PMID 12973660
- [Background] Krupp LB, Tardieu M, Amato MP, Banwell B, Chitnis T, Dale RC, Ghezzi A, Hintzen R, Kornberg A, Pohl D, Rostasy K, Tenembaum S, Wassmer E; International Pediatric Multiple Sclerosis Study Group. International Pediatric Multiple Sclerosis Study Group criteria for pediatric multiple sclerosis and immune-mediated central nervous system demyelinating disorders: revisions to the 2007 definitions. Mult Scler. 2013 Sep;19(10):1261-7. doi: 10.1177/1352458513484547. Epub 2013 Apr 9. PMID 23572237
- [Background] Verhey LH, Branson HM, Shroff MM, Callen DJ, Sled JG, Narayanan S, Sadovnick AD, Bar-Or A, Arnold DL, Marrie RA, Banwell B; Canadian Pediatric Demyelinating Disease Network. MRI parameters for prediction of multiple sclerosis diagnosis in children with acute CNS demyelination: a prospective national cohort study. Lancet Neurol. 2011 Dec;10(12):1065-73. doi: 10.1016/S1474-4422(11)70250-2. Epub 2011 Nov 6. PMID 22067635
- [Background] Pohl D, Alper G, Van Haren K, Kornberg AJ, Lucchinetti CF, Tenembaum S, Belman AL. Acute disseminated encephalomyelitis: Updates on an inflammatory CNS syndrome. Neurology. 2016 Aug 30;87(9 Suppl 2):S38-45. doi: 10.1212/WNL.0000000000002825. PMID 27572859